CLINICAL TRIAL: NCT03633058
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over Study to Assess the Safety, Tolerability and Efficacy of Oral Ketamine for Patients With Rett Syndrome
Brief Title: A Study to Evaluate Ketamine for the Treatment of Rett Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rett Syndrome Research Trust (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Neul, Director, Vanderbilt Kennedy Center, Annette Schaffer Eskind Chair, Professor of Pediatrics, Pharmacology, and Special Education, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Ket-101-RSRT
Record Dates: First submitted 2018-08-08; First posted 2018-08-16 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Rett Syndrome
Keywords: MECP2; RTT; Retts; ketamine
MeSH Terms: conditions — Rett Syndrome | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Patients will receive placebo and ketamine for 5 days BID each, in a double-blind treatment order, and will be assessed for 2 weeks after each treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.75 mg/kg (Experimental): ketamine will be dosed orally twice daily for 5 days at 0.75 mg/kg, in addition to 5 days of placebo
  Interventions: Drug: Ketamine
- 1.5 mg/kg (Experimental): ketamine will be dosed orally twice daily for 5 days at 0.75 mg/kg, in addition to 5 days of placebo
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — oral ketamine dosed twice daily for 5 days
  Other Names: Ketalar

SUMMARY:
This 2 cohort, sequential, ascending dose study will assess the safety, tolerability and efficacy of oral ketamine dosed in a single 5-day BID regimen in addition to placebo, in a 4-week cross-over design in patients with Rett Syndrome. Approximately 12 patients per cohort are anticipated to participate for approximately 8-10 weeks at approximately 7 US study centers.

DETAILED DESCRIPTION:
This study is designed to assess oral ketamine for the treatment of Rett Syndrome and consists of up to 4 ascending dose cohorts, each assessing 1 dose level of ketamine vs placebo. Patients will receive in either order, a 5-day BID regimen of both placebo and the cohort-specified dose level of oral ketamine. Patients may only participate in 1 cohort. Safety and tolerability will be assessed via patient disposition, vital signs, physical examination, adverse events and concomitant medication use. Efficacy will be assessed via physician and caregiver questionnaires and assessments, and continuous, wearable, at-home biosensor data collection. An independent safety committee will review safety data from each cohort to determine if the subsequent ascending dose cohort is warranted. A total of 12 patients per cohort is anticipated at approximately 7 sites. The screening period will last between 2 and 4 weeks, the cross-over treatment period will last 4 weeks, and the safety follow-up period will last 2 weeks. Total patient participation is approximately 8-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female Rett Syndrome patients diagnosed with Rett Syndrome with a confirmed MECP2 mutation
* between the ages of 6 and 12, inclusive, who have not achieved menarche
* ability to take oral medications
* are generally healthy.

Exclusion Criteria:

* Patients not on stable medication regimens/other types of behavioral, educational, or dietary interventions for at least 4 weeks,
* are taking medications that may interact with ketamine,
* have a condition where increased blood pressure, spinal fluid pressure, or ocular pressure may put the patient at increased risk.

Ages: 6 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Neul, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Jana von Hehn, PhD, Study Director — Rett Syndrome Research Trust
Locations (7):
- United States (7):
  - University of Alabama Birmingham School of Medicine, Birmingham, Alabama
  - Children's Hospital Colorado, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campbell K, Neul JL, Lieberman DN, Berry-Kravis E, Benke TA, Fu C, Percy A, Suter B, Morris D, Carpenter RL, Marsh ED, von Hehn J. A randomized, placebo-controlled, cross-over trial of ketamine in Rett syndrome. J Neurodev Disord. 2025 Jan 24;17(1):4. doi: 10.1186/s11689-025-09591-y. PMID 39856538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 sites in the US with active participants between 12Mar2019 and 22Nov2021.
Pre-assignment Details: 24 participants were screened, 23 were enrolled. 23 patients were included in the safety analysis. 21 were included in the efficacy analysis (1 was withdrawn, and 1 was excluded from analysis for study ineligibility).
Groups:
- 0.75 mg/kg (Placebo First, Then 0.75 mg/kg Ketamine); 1.5 mg/kg (Placebo First, Then 1.5 mg/kg Ketamine): placebo was dosed orally twice daily for 5 days followed by ketamine dosed orally twice daily for 5 days at 0.75 mg/kg. Dosing initiations were 14 days apart.
- 0.75 mg/kg (0.75 mg/kg Ketamine First, Then Placebo): ketamine was dosed orally twice daily for 5 days at 0.75 mg/kg followed by placebo dosed orally twice daily for 5 days. Dosing initiations were 14 days apart.
- 1.5 mg/kg (1.5 mg/kg Ketamine First, Then Placebo): ketamine was dosed orally twice daily for 5 days at 1.5 mg/kg followed by placebo dosed orally twice daily for 5 days. Dosing initiations were 14 days apart.
Period: Overall Study
Arm/Group | 0.75 mg/kg (Placebo First, Then 0.75 mg/kg Ketamine) | 0.75 mg/kg (0.75 mg/kg Ketamine First, Then Placebo) | 1.5 mg/kg (Placebo First, Then 1.5 mg/kg Ketamine) | 1.5 mg/kg (1.5 mg/kg Ketamine First, Then Placebo)
Started | 5 | 6 | 6 | 6
Completed | 5 | 6 | 5 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants - 0.75 mg/kg Ketamine; All Study Participants - 1.5 mg/kg Ketamine: Female patients with Rett syndrome, aged 6-12 years inclusive, who had not achieved menarche.
- Total: Total of all reporting groups
Arm/Group | All Study Participants - 0.75 mg/kg Ketamine | All Study Participants - 1.5 mg/kg Ketamine | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (2.20) | 7.6 (1.93) | 8.1 (2.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 11 | 20
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23
Weight [Mean (Standard Deviation); unit: kg] | 24.4 (7.33) | 21.5 (4.62) | 22.9 (6.10)
Height [Mean (Standard Deviation); unit: cm] — Population: 1 pt was not measured for height
  cm
    number analyzed (Participants) | 11 | 11 | 22
    (all) | 126.0 (11.84) | 117.5 (9.41) | 121.7 (11.30)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: 1 pt was not measured for height and BMI could not be calculated
  kg/m^2
    number analyzed (Participants) | 11 | 11 | 22
    (all) | 15.1 (3.06) | 15.4 (1.89) | 15.2 (2.48)

OUTCOME MEASURES:

1. Primary Outcome: Dose-Limiting Adverse Events
Description: The Number of Participants with Treatment-emergent adverse events on ketamine compared to placebo will be summarized
Time Frame: 6 weeks
Population: The Safety Population consisted of all patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- 0.75 mg/kg Ketamine: ketamine was dosed orally twice daily for 5 days at 0.75 mg/kg and placebo was dosed orally twice daily for 5 days. Dose initiations were 14 days apart. AEs reported occurred while patients were on ketamine.
- 0.75 mg/kg Placebo: placebo was dosed orally twice daily for 5 days and ketamine was dosed orally at 0.75 mg/kg twice daily for 5 days. Dose initiations were 14 days apart. AEs reported occurred while patients were on placebo.
- 1.5 mg/kg Ketamine: ketamine was dosed orally twice daily for 5 days at 1.5 mg/kg and placebo was dosed orally twice daily for 5 days. Dose initiations were 14 days apart. AEs reported occurred while patients were on ketamine.
- 1.5 mg/kg Placebo: placebo was dosed orally twice daily for 5 days and ketamine was dosed orally at 1.5 mg/kg twice daily for 5 days. Dose initiations were 14 days apart. AEs reported occurred while patients were on placebo.
Arm/Group | 0.75 mg/kg Ketamine | 0.75 mg/kg Placebo | 1.5 mg/kg Ketamine | 1.5 mg/kg Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
Participants
  TEAEs | 2 | 4 | 6 | 3
  SAEs | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 0 | 1 | 0
  AEs leading to dose interruption | 0 | 0 | 0 | 0
  No TEAEs reported | 9 | 7 | 5 | 9

2. Other Pre Specified Outcome: Continuous Biosensor Data
Description: 2 different non-invasive, wearable devices will be used in the study to determine changes in physiologic measures for the patient in the home environment. Biosensors will be worn continuously during the screening and treatment period to measure activity, sleep, position, heart rate, and breathing.
Time Frame: 6-8 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Clinical Global Impression of Improvement
Description: Clinicians will use a 7 point Likert Scale to rate change from baseline symptom severity by addressing the question, "Compared to the patient's condition of Rett syndrome prior to treatment initiation at baseline, the patient's current condition is: 1 very much improved, 2 much improved, 3 minimally improved, 4 no change, 5 minimally worse, 6 much worse, 7 very much worse. No change would be scored a 0, while improvement would be scored at -1, -2, or -3 and worsening would be scored +1, +2 or +3, depending on the degree of perceived change. Negative change indicates improvement while positive change indicates worsening
Time Frame: 4 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Motor Behavioral Assessment
Description: a 37-item questionnaire for clinicians to evaluate current behavioral/social, orofacial/respiratory, and motor/physical symptoms. Each item is rated either 0 (normal or never), 1 (mild or rare), 2 (moderate or occasional), 3 (marked or frequent), 4 (very severe or constant), where higher numbers indicate higher severity. Each subscale is summed for a subscale score, while the total score is a sum of the subscale scores. The behavioral/social subscale score may range from 0 to 64; the orofacial/respiratory subscale may range from 0 to 28, and motor/physical subscale may range from 0 to 56. Total score may range from 0 to 148.
Time Frame: 4 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Clinician Domain Likert Scale
Description: an 8 category (domain) questionnaire to assess current hand function, walking, verbal and non-verbal communication, comprehension, attention, behavior problems, and mood by considering the question, "Considering your experience with the patient at this visit, please rate the level of function in each category". Each domain will be rated on a 7 point Likert Scale where the clinician will select 1 of 7 choices: 1 normal, 2 borderline abnormal, 3 mildly abnormal, 4 moderately abnormal, 5 markedly abnormal, 6 severely abnormal, 7 extremely abnormal. Lower values indicate lesser severity while higher values indicate higher severity.
Time Frame: 4 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Rett Syndrome Behaviour Questionnaire
Description: a 45-item questionnaire for clinicians to evaluate current behavior and emotional features. Each item is rated either 0 (not true or not done), 1 (somewhat or sometimes true) and 2 (very true), where higher numbers indicate higher severity. Total score is summed and may range from 0 to 90.
Time Frame: 4 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Parent Domain Likert Scale
Description: a 9 category (domain) questionnaire to assess current hand function, walking, verbal and non-verbal communication, comprehension, attention, behavior problems, mood, and seizure activity, by considering the question, "Considering your experience with your child over the past 7 days, please rate your child's level of function in each category". Each domain will be rated on a 7 point Likert Scale where the parent/caregiver will select 1 of 7 choices: 1 normal, 2 borderline abnormal, 3 mildly abnormal, 4 moderately abnormal, 5 markedly abnormal, 6 severely abnormal, 7 extremely abnormal. Lower values indicate lesser severity while higher values indicate higher severity.
Time Frame: 4 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Children's Sleep Habits Questionnaire
Description: a 35-item questionnaire for parents to evaluate current sleep and common sleep problems. The parent/caregiver will rate each item as 1 (rarely), 2 (sometimes), or 3 (usually), where higher scores indicate higher severity. The parent/caregiver will also indicate if the item is a problem or not. A total score of the sum of each item and 8 subscale scores (bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep disordered breathing, and daytime sleepiness) are possible. Total scores between 0 and 70 are possible, where higher scores indicate more sleep problems.
Time Frame: 4 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Rett Caregiver Burden Inventory Assessment
Description: a 26-item questionnaire for parents to evaluate the burden of care on their quality of life. The parent/caregiver will rate each item as 0 (never), 1 (rarely), 2 (sometimes), 3 (quite frequently), or 4 (nearly always) where higher scores indicate higher severity. Total scores between 0 and 104 are possible, where higher scores indicate more caregiver burden.
Time Frame: 4 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: EEG Signature
Description: ketamine EEG alpha, beta, gamma, delta and theta waveform signatures compared to placebo to indicate target engagement
Time Frame: Day 1, Day 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- 0.75 mg/kg Ketamine: AEs reported while on ketamine in the 0.75 mg/kg cohort
- 0.75 mg/kg Placebo: AEs reported while on placebo in the 0.75 mg/kg cohort
- 1.5 mg/kg Ketamine: AEs reported while on ketamine in the 1.5 mg/kg cohort
- 1.5 mg/kg Placebo: AEs reported while on placebo in the 1.5 mg/kg cohort
Arm/Group | 0.75 mg/kg Ketamine | 0.75 mg/kg Placebo | 1.5 mg/kg Ketamine | 1.5 mg/kg Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/11 | 4/11 | 7/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 4.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.75 mg/kg Ketamine (N=11) | 0.75 mg/kg Placebo (N=11) | 1.5 mg/kg Ketamine (N=12) | 1.5 mg/kg Placebo (N=12)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma site irritation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
sedation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonic convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT03633058/Prot_SAP_000.pdf